CLINICAL TRIAL: NCT02909426
Title: Effectiveness of Breast Cancer Screening in Women Aged 40-59: Digital Mammography With Supplemental Breast Ultrasonography Versus Digital Mammography Only
Brief Title: The Mammography and Ultrasonography STudy for Breast Cancer Screening Effectiveness
Acronym: MUST-BE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, EUN HYE LEE, Director, Head of Breast Imaging, Principal Investigator, Professor, Soonchunhyang University Hospital
Other Study IDs: 1520200
Record Dates: First submitted 2016-09-05; First posted 2016-09-21 (Estimated); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Invasive Cancer; Ductal Carcinoma in Situ
Keywords: Screening; Digital mammography; Ultrasonography; Sensitivity; Specificity
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Hypersensitivity | interventions — Ultrasonography; Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women aged 40-59: Asymptomatic women aged 40-59 who participate in the National Cancer Screening Program in Korea and agreed with participating in this study will be the cohort.
  The participants' digital mammography and ultrasonography will be interpreted combinedly by radiologists who perform the screening sonography and the participants' digital mammography will be interpreted independently by other radiologists who do not perform the screening sonography.
  Interventions: Device: Ultrasonography; Device: Digital mammography

INTERVENTIONS:
Device: Ultrasonography — Radiologists' hand-held bilateral breast ultrasonography for each participant for one time
Device: Digital mammography — Full-field digital mammography using one of the equipments from General Electric (GE), Hologic, and Medi-future companies for each participant for one time

SUMMARY:
Mammography screening has limited performance in young women or women with dense breasts although it is the only proven method for breast cancer screening that reduces the mortality. The investigators propose a multicenter trial of breast cancer screening to assess the effectiveness of supplemental ultrasonography for Korean women aged 40-59 years.

DETAILED DESCRIPTION:
The investigators will screen same consecutive participants using both methods; digital mammography plus supplemental ultrasonography (intervention arm) and digital mammography only (control arm) for 5 years. The investigators will collect follow-up information by assessment of screening records, questionnaire, and official cancer registry. The primary outcome will be sensitivity, specificity, recall rate, cancer detection rate and stage distribution at the end of first round of screening. The secondary outcome will be cost-effectiveness and cost-utility of digital mammography with ultrasonography versus digital mammography only for breast cancer screening. It is hoped that the results of this trial will provide guidance of effective breast cancer screening strategy to women aged 40-59, especially with dense breasts.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-59 years
* No history of any cancer
* No breast mammography (and ultrasonography, in case of intervention arm) after the introduction of digital mammography

Exclusion Criteria:

* Interstitial injection
* Women with history of any cancer

Ages: 40 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 40-59 years at target population in National Cancer Screening Program
Sampling Method: Non-Probability Sample
Enrollment: 11880 (Actual)
Dates: Start 2016-05-02 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of digital mammography with supplemental breast ultrasonography and digital mammography only | 1 year after the screening
  rate of positive results of the screening among histologically proved breast cancer patients

SECONDARY OUTCOMES:
Cost-effectiveness of supplemental ultrasonography of the breast | 1 year after the screening
  Comparison of the cost for detecting one breast cancer patient by two groups.
Cost-utility of supplemental ultrasonography of the breast | 1 year after the screening
  Measurement of the incremental cost-utility ratio, which is calculated by dividing the difference in costs by difference in the quality-adjusted life year (QALY).

CONTACTS AND LOCATIONS:
Overall Officials: EUN HYE LEE, MD, Ph.D, Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Soon Chun Hyang University Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohuchi N, Suzuki A, Sobue T, Kawai M, Yamamoto S, Zheng YF, Shiono YN, Saito H, Kuriyama S, Tohno E, Endo T, Fukao A, Tsuji I, Yamaguchi T, Ohashi Y, Fukuda M, Ishida T; J-START investigator groups. Sensitivity and specificity of mammography and adjunctive ultrasonography to screen for breast cancer in the Japan Strategic Anti-cancer Randomized Trial (J-START): a randomised controlled trial. Lancet. 2016 Jan 23;387(10016):341-348. doi: 10.1016/S0140-6736(15)00774-6. Epub 2015 Nov 5. PMID 26547101